CLINICAL TRIAL: NCT02896400
Title: Optimizing Tobacco Dependence Treatment in the Emergency Department
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1603017332; 1R01CA201873-01A1 (NIH)
Record Dates: First submitted 2016-09-06; First posted 2016-09-12 (Estimated); Results first posted 2020-11-16 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (16):
- BNI+NRT+QL+Text (Experimental): Brief Negotiated Interview (BNI) Nicotine replacement therapy (NRT) patches and gum, 6 weeks supply Referral to CT Smokers Quitline (QL) Registration in SmokefreeText (Text)
  Interventions: Behavioral: Brief Negotiated Interview (BNI); Drug: Nicotine replacement therapy (NRT); Other: CT Smokers Quitline (QL); Other: SmokefreeText (Text)
- BNI+NRT+QL (Experimental): Brief Negotiated Interview (BNI) Nicotine replacement therapy (NRT) patches and gum, 6 weeks supply Referral to CT Smokers Quitline (QL)
  Interventions: Behavioral: Brief Negotiated Interview (BNI); Drug: Nicotine replacement therapy (NRT); Other: CT Smokers Quitline (QL)
- BNI+NRT+Text (Experimental): Brief Negotiated Interview (BNI) Nicotine replacement therapy (NRT) patches and gum, 6 weeks supply Registration in SmokefreeText (Text)
  Interventions: Behavioral: Brief Negotiated Interview (BNI); Drug: Nicotine replacement therapy (NRT); Other: SmokefreeText (Text)
- BNI+NRT (Experimental): Brief Negotiated Interview (BNI) Nicotine replacement therapy (NRT) patches and gum, 6 weeks supply
  Interventions: Behavioral: Brief Negotiated Interview (BNI); Drug: Nicotine replacement therapy (NRT)
- BNI+QL+Text (Experimental): Brief Negotiated Interview (BNI) Referral to CT Smokers Quitline (QL) Registration in SmokefreeText (Text)
  Interventions: Behavioral: Brief Negotiated Interview (BNI); Other: CT Smokers Quitline (QL); Other: SmokefreeText (Text)
- BNI+QL (Experimental): Brief Negotiated Interview (BNI) Referral to CT Smokers Quitline (QL)
  Interventions: Behavioral: Brief Negotiated Interview (BNI); Other: CT Smokers Quitline (QL)
- BNI+Text (Experimental): Brief Negotiated Interview (BNI) Registration in SmokefreeText (Text)
  Interventions: Behavioral: Brief Negotiated Interview (BNI); Other: SmokefreeText (Text)
- BNI only (Experimental): Brief Negotiated Interview (BNI)
  Interventions: Behavioral: Brief Negotiated Interview (BNI)
- NRT+QL+Text (Experimental): Nicotine replacement therapy (NRT) patches and gum, 6 weeks supply Referral to CT Smokers Quitline (QL) Registration in SmokefreeText (Text)
  Interventions: Drug: Nicotine replacement therapy (NRT); Other: CT Smokers Quitline (QL); Other: SmokefreeText (Text)
- NRT+QL (Experimental): Nicotine replacement therapy (NRT) patches and gum, 6 weeks supply Referral to CT Smokers Quitline (QL)
  Interventions: Drug: Nicotine replacement therapy (NRT); Other: CT Smokers Quitline (QL)
- NRT+Text (Experimental): Nicotine replacement therapy (NRT) patches and gum, 6 weeks supply Registration in SmokefreeText (Text)
  Interventions: Drug: Nicotine replacement therapy (NRT); Other: SmokefreeText (Text)
- NRT only (Experimental): Nicotine replacement therapy (NRT) patches and gum, 6 weeks supply
  Interventions: Drug: Nicotine replacement therapy (NRT)
- QL+Text (Experimental): Referral to CT Smokers Quitline (QL) Registration in SmokefreeText (Text)
  Interventions: Other: CT Smokers Quitline (QL); Other: SmokefreeText (Text)
- QL only (Experimental): Referral to CT Smokers Quitline (QL)
  Interventions: Other: CT Smokers Quitline (QL)
- Text only (Experimental): Registration in SmokefreeText (Text)
  Interventions: Other: SmokefreeText (Text)
- Control (No Intervention): Control arm, no intervention

INTERVENTIONS:
Behavioral: Brief Negotiated Interview (BNI) — Brief motivational interview on smoking behavior
  Arms: BNI only; BNI+NRT; BNI+NRT+QL; BNI+NRT+QL+Text; BNI+NRT+Text; BNI+QL; BNI+QL+Text; BNI+Text
Drug: Nicotine replacement therapy (NRT) — 6 weeks of nicotine replacement, patches and gum. First dose of each started in ED. Patches are 14mg or 21 mg. Gum is 2mg per piece.
  Arms: BNI+NRT; BNI+NRT+QL; BNI+NRT+QL+Text; BNI+NRT+Text; NRT only; NRT+QL; NRT+QL+Text; NRT+Text
Other: CT Smokers Quitline (QL) — Faxed referral to the CT Smokers Quitline for the subject. QL will then call subject to offer phone based counseling.
  Arms: BNI+NRT+QL; BNI+NRT+QL+Text; BNI+QL; BNI+QL+Text; NRT+QL; NRT+QL+Text; QL only; QL+Text
Other: SmokefreeText (Text) — Enrollment in a version of NCI's SmokefreeTxt, tailored for the study.
  Arms: BNI+NRT+QL+Text; BNI+NRT+Text; BNI+QL+Text; BNI+Text; NRT+QL+Text; NRT+Text; QL+Text; Text only

SUMMARY:
The investigators propose an innovative full-factorial design in a cohort of 1056 adult smokers in an urban emergency department (ED), to test the efficacy of four key intervention components: motivational interviewing, medication, quitline referral, and texting. At the trial's completion, a mixed-methods approach will be used to identify the components that were efficacious within the proposed cost constraint, along with feasibility and acceptability to providers and subjects. The investigators will then assemble an intervention that maximizes efficacy, given a cost-effectiveness constraint and findings from a qualitative analysis.

DETAILED DESCRIPTION:
The investigators propose to optimize the identification and treatment of adult smokers seen in a hospital ED. To do this the Multiple Optimization Strategy (MOST) will be employed to develop a multicomponent intervention that will consist of some combination of the following: (1) a Brief Negotiation Interview (BNI, a variant of a motivational interview), delivered by a trained research assistant; (2) provision of 6 weeks of nicotine patches and gum to the research participant, with application of the first patch in the ED (NRT); (3) active referral to the Connecticut Smokers' Quitline (QL); and (4) enrollment in the SmokefreeText a short-messaging service (SMS) texting program for mobile phones (Text). Using MOST principles, the first phase of the study will use a 2x2x2x2 full-factorial design to identify the components most likely to be efficacious in combination. Although the factorial design requires the allocation of participants to 16 different combinations of the 4 components (Table 1), evaluation of each individual component is performed comparing all of those receiving a component to all of those not receiving a component, making this an efficient design. For instance, evaluation of the BNI component will compare those randomized to arms 1 through 8 to those in arms 9 to 16.The second phase will consist of designing and proposing a 2-arm randomized clinical trial comparing the efficacy of the multicomponent intervention package to usual care; this will be conducted in a future application.

The specific aims of this proposed study are:

Aim 1. To conduct a fully powered factorial randomized trial of 1056 adult smokers to test the efficacy of 4 key components of ED-initiated tobacco treatment: Brief Negotiated Interview (BNI), nicotine replacement therapy (NRT), Quitline referral (QL), and SmokeFreeText (Text).

Aim 2. To identify the most efficacious components of our intervention, within fixed constraints of cost effectiveness and feasibility/acceptability to providers and subjects.

Aim 3. To lay the groundwork for a future randomized trial testing the previously identified components, delivered as a package, against a control arm in a new cohort of adult ED smokers.

Our associated hypotheses are:

1. At 3 months, at least 1 intervention component will yield a biochemically verified tobacco abstinence rate at least 5% greater than in the control condition. Carbon monoxide breath test will be used for biochemical verification.
2. At 3 months, at least 1 intervention will be cost-effective, using a societal perspective.
3. At 3 months, at least 1 intervention will be acceptable and feasible to providers and subjects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* have smoked >= 100 cigarettes lifetime
* describe themselves as every or some day smokers
* smoke at least 5 cigarettes/day
* own a cellphone with texting capability
* are able to give written informed consent

Exclusion Criteria:

* Inability to read or understand English
* currently receiving formal tobacco dependence treatment
* life-threatening or unstable medical, surgical, or psychobehavioral condition
* unable to provide at least one collateral contact
* live out-of-state
* leaving the ED against medical advice
* pregnant (self-report or urine testing), nursing, or trying to conceive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1056 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Bernstein, MD, Principal Investigator — Yale School of Medicine, Department of Emergency Medicine
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bernstein SL, Dziura J, Weiss J, Miller T, Vickerman KA, Grau LE, Pantalon MV, Abroms L, Collins LM, Toll B. Tobacco dependence treatment in the emergency department: A randomized trial using the Multiphase Optimization Strategy. Contemp Clin Trials. 2018 Mar;66:1-8. doi: 10.1016/j.cct.2017.12.016. Epub 2017 Dec 27. PMID 29287665

RESULTS

PARTICIPANT FLOW:
Period: Baseline
Arm/Group | NRT+QL+Text | BNI+QL+Text | BNI+NRT+QL+Text | NRT+QL | BNI+QL | NRT Only | BNI+Text | BNI+NRT+Text | NRT+Text | BNI+NRT | Control | BNI+NRT+QL | Text Only | QL+Text | BNI Only | QL Only
Started | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66
Completed | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: 1 Month Follow-up
Arm/Group | NRT+QL+Text | BNI+QL+Text | BNI+NRT+QL+Text | NRT+QL | BNI+QL | NRT Only | BNI+Text | BNI+NRT+Text | NRT+Text | BNI+NRT | Control | BNI+NRT+QL | Text Only | QL+Text | BNI Only | QL Only
Started | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66
Completed | 59 | 59 | 61 | 58 | 57 | 60 | 61 | 60 | 62 | 59 | 61 | 61 | 63 | 62 | 65 | 63
Not Completed | 7 | 7 | 5 | 8 | 9 | 6 | 5 | 6 | 4 | 7 | 5 | 5 | 3 | 4 | 1 | 3
Not completed — Lost to Follow-up | 7 | 7 | 5 | 8 | 9 | 6 | 5 | 6 | 4 | 7 | 5 | 5 | 3 | 4 | 1 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: 3 Month Follow-up
Arm/Group | NRT+QL+Text | BNI+QL+Text | BNI+NRT+QL+Text | NRT+QL | BNI+QL | NRT Only | BNI+Text | BNI+NRT+Text | NRT+Text | BNI+NRT | Control | BNI+NRT+QL | Text Only | QL+Text | BNI Only | QL Only
Started (We call all participants at the 3m follow-up time point even if the 1m follow-up was not completed.) | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 65
Completed | 60 | 63 | 60 | 55 | 54 | 60 | 62 | 63 | 60 | 61 | 60 | 60 | 63 | 60 | 62 | 63
Not Completed | 6 | 3 | 6 | 11 | 12 | 6 | 4 | 3 | 6 | 5 | 6 | 6 | 3 | 6 | 4 | 2
Not completed — Lost to Follow-up | 6 | 3 | 6 | 11 | 12 | 6 | 4 | 3 | 6 | 5 | 6 | 6 | 3 | 5 | 3 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Period: Biochemical Verification at 3 Months
Arm/Group | NRT+QL+Text | BNI+QL+Text | BNI+NRT+QL+Text | NRT+QL | BNI+QL | NRT Only | BNI+Text | BNI+NRT+Text | NRT+Text | BNI+NRT | Control | BNI+NRT+QL | Text Only | QL+Text | BNI Only | QL Only
Started | 60 | 63 | 60 | 55 | 54 | 60 | 62 | 63 | 60 | 61 | 60 | 60 | 63 | 60 | 62 | 63
Completed (Only participants reporting abstinence at the 3m follow-up complete the biochem.) | 14 | 15 | 13 | 14 | 9 | 11 | 11 | 14 | 15 | 8 | 5 | 19 | 10 | 12 | 7 | 6
Not Completed | 46 | 48 | 47 | 41 | 45 | 49 | 51 | 49 | 45 | 53 | 55 | 41 | 53 | 48 | 55 | 57
Not completed — Lost to Follow-up | 1 | 0 | 1 | 1 | 0 | 1 | 3 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 3 | 1
Not completed — participant was not eligible for biochem | 45 | 48 | 46 | 40 | 45 | 48 | 48 | 47 | 44 | 52 | 55 | 41 | 52 | 48 | 52 | 56

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NRT+QL+Text | BNI+QL+Text | BNI+NRT+QL+Text | NRT+QL | BNI+QL | NRT Only | BNI+Text | BNI+NRT+Text | NRT+Text | BNI+NRT | Control | BNI+NRT+QL | Text Only | QL+Text | BNI Only | QL Only | Total
Number analyzed (Participants) | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 1056
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.86 (10.72) | 41.33 (11.92) | 44.36 (12.75) | 43.73 (12.14) | 40.56 (11.97) | 42.26 (12.27) | 42.64 (12.42) | 43.77 (11.80) | 43.67 (12.60) | 44.30 (13.23) | 43.65 (14.00) | 43.18 (10.67) | 44.33 (12.23) | 42.36 (12.49) | 41.86 (10.42) | 43.21 (11.77) | 43.26 (12.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 38 | 35 | 28 | 28 | 31 | 34 | 28 | 41 | 35 | 35 | 29 | 33 | 42 | 31 | 36 | 536
  Male | 34 | 28 | 31 | 38 | 38 | 35 | 32 | 38 | 25 | 31 | 31 | 37 | 33 | 24 | 35 | 30 | 520
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 15 | 7 | 22 | 15 | 9 | 19 | 10 | 14 | 23 | 13 | 14 | 13 | 19 | 14 | 10 | 231
  Not Hispanic or Latino | 52 | 51 | 56 | 43 | 51 | 55 | 45 | 55 | 51 | 43 | 52 | 49 | 51 | 45 | 52 | 56 | 807
  Unknown or Not Reported | 0 | 0 | 3 | 1 | 0 | 2 | 2 | 1 | 1 | 0 | 1 | 3 | 2 | 2 | 0 | 0 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 1 | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 15
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 9
  Black or African American | 24 | 25 | 34 | 22 | 26 | 24 | 23 | 23 | 23 | 19 | 27 | 26 | 29 | 28 | 19 | 29 | 401
  White | 39 | 33 | 26 | 35 | 33 | 36 | 36 | 35 | 37 | 40 | 29 | 35 | 30 | 28 | 34 | 31 | 537
  More than one race | 0 | 5 | 3 | 5 | 2 | 6 | 4 | 5 | 2 | 5 | 7 | 0 | 2 | 5 | 10 | 2 | 63
  Unknown or Not Reported | 0 | 1 | 2 | 3 | 2 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 5 | 4 | 2 | 3 | 28
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 66 | 1056
Cigarettes per Day (CPD) [Median (Inter-Quartile Range); unit: cigarettes per day] — Number of cigarettes smoked per day at baseline
  cigarettes per day | 10.0 [7 to 15] | 12.0 [8 to 20] | 10.0 [6 to 12] | 10.0 [6 to 13] | 10.0 [5 to 15] | 10.0 [6 to 12] | 10.0 [6 to 15] | 10.0 [5 to 15] | 9.0 [5 to 15] | 10.0 [7 to 20] | 10.0 [5 to 15] | 11.0 [7 to 20] | 10.0 [8 to 15] | 10.0 [5 to 15] | 10.0 [6 to 15] | 10.0 [6 to 15] | 10.0 [5 to 20]
Heaviness of Smoking Index >=4 [Number; unit: participants] — Heaviness of Smoking Index score derived from 2 questions:
  1. On the days that you smoke, how soon after you wake up do you have your first cigarette?
  2. How many cigarettes do you typically smoke per day?
  SCORING:
  0-2: low addiction 3-4: moderate addiction 5-6: high addiction
  participants | 15 | 28 | 13 | 18 | 9 | 23 | 20 | 13 | 13 | 21 | 15 | 21 | 19 | 13 | 17 | 12 | 270

OUTCOME MEASURES:

1. Primary Outcome: Tobacco Abstinence
Description: Abstinence self reported and verified by exhaled carbon monoxide
Time Frame: 3 months
Population: All participants eligible for 3 month follow-up (deceased participants excluded). Each intervention group was compared with all participants who did not receive that intervention. The comparison group therefore differed for each intervention: BNI=526; NRT=525; QL=527; Text = 526.
Measure: Count of Participants; unit: Participants
Groups:
- Brief Negotiated Interview (BNI): All 8 arms with Brief Negotiated Interview as an intervention:
  BNI only BNI+Nicotine Replacement Therapy (NRT) BNI+Quitline (QL) BNI+Text BNI+NRT+QL BNI+NRT+Text BNI+QL+Text BNI+NRT+QL+Text
- Brief Negotiated Interview (BNI) CONTROL: All 8 arms which did not include the BNI intervention:
  NRT+QL+Text NRT+QL NRT+Text NRT QL+Text QL Text Control
- Nicotine Replacement Therapy (NRT): All 8 arms with Nicotine Replacement Therapy as an intervention:
  NRT only Brief Negotiated Interview (BNI)+NRT NRT+Quitline (QL) NRT+Text BNI+NRT+QL BNI+NRT+Text NRT+QL+Text BNI+NRT+QL+Text
- Nicotine Replacement Therapy (NRT) CONTROL: All 8 arms which did not include the NRT intervention:
  BNI+QL+Text BNI+QL BNI+Text BNI Only QL+Text QL Only Text Only Control
- Quitline (QL): All 8 arms with the Quitline as an intervention:
  QL only Brief Negotiated Interview (BNI)+QL Nicotine Replacement Therapy (NRT)+QL QL+Text BNI+NRT+QL BNI+QL+Text NRT+QL+Text BNI+NRT+QL+Text
- Quitline (QL) CONTROL: All 8 arms which did not include the QL intervention:
  BNI+NRT+Text BNI+NRT BNI+Text BNI Only NRT+Text NRT Only Text Only Control
- Text: All 8 arms with Text as an intervention:
  Text only Brief Negotiated Interview (BNI)+Text Nicotine Replacement Therapy (NRT)+Text Quitline (QL)+Text BNI+NRT+Text BNI+QL+Text NRT+QL+Text BNI+NRT+QL+Text
- Text CONTROL: All 8 arms which did not include the Text intervention:
  BNI+NRT+QL BNI+NRT BNI+QL BNI Only NRT+QL NRT Only QL Only Control
Arm/Group | Brief Negotiated Interview (BNI) | Brief Negotiated Interview (BNI) CONTROL | Nicotine Replacement Therapy (NRT) | Nicotine Replacement Therapy (NRT) CONTROL | Quitline (QL) | Quitline (QL) CONTROL | Text | Text CONTROL
Number analyzed (Participants) | 527 | 526 | 528 | 525 | 526 | 527 | 527 | 526
Participants | 71 | 49 | 76 | 44 | 66 | 54 | 61 | 59
Statistical Analysis 1: Comparison: Brief Negotiated Interview (BNI) vs Brief Negotiated Interview (BNI) CONTROL; 8 arms including BNI (BNI only, BNI+NRT, BNI+QL, BNI+Text, BNI+NRT+QL, BNI+NRT+Text, BNI+QL+Text, BNI+NRT+QL+Text) compared to the 8 arms that do not include BNI (Control, NRT only, QL only, Text only, NRT+QL, NRT+Text, QL+Text, NRT+QL+Text); Test type: Superiority; p = .01, Regression, Logistic; Adjusted for gender, age, race/ethnicity, baseline daily cigarette consumption; Odds Ratio (OR) = 1.8, 95% CI 2-sided [1.1 to 2.8]
Statistical Analysis 2: Comparison: Nicotine Replacement Therapy (NRT) vs Nicotine Replacement Therapy (NRT) CONTROL; 8 arms that include NRT (NRT only, BNI+NRT, NRT+QL, NRT+Text, BNI+NRT+QL, BNI+NRT+Text, NRT+QL+Text, BNI+NRT+QL+Text) compared to 8 arms that do not include NRT (Control, BNI only, QL only, Text only, BNI+QL, BNI+Text, QL+Text, BNI+QL+Text); Test type: Superiority; p = .001, Regression, Logistic; adjusted for gender, age, race/ethnicity, baseline daily cigarette consumption; Odds Ratio (OR) = 2.1, 95% CI 2-sided [1.3 to 3.2]
Statistical Analysis 3: Comparison: Quitline (QL) vs Quitline (QL) CONTROL; 8 arms including QL intervention (QL only, BNI+QL, NRT+QL, QL+Text, BNI+NRT+QL, BNI+QL+Text, NRT+QL+Text, BNI+NRT+QL+Text) compared to all 8 arms that did not include QL (Control, BNI only, NRT only, Text only, BNI+NRT, BNI+Text, NRT+Text, BNI+NRT+Text); Test type: Superiority; p = 0.14, Regression, Logistic; adjusted for gender, age, race/ethnicity, baseline daily cigarette consumption; Odds Ratio (OR) = 1.4, 95% CI 2-sided [0.9 to 2.2]
Statistical Analysis 4: Comparison: Text vs Text CONTROL; 8 arms including Text (Text only, BNI+Text, NRT+Text, QL+Text, BNI+NRT+Text, BNI+QL+Text, NRT+QL+Text, BNI+NRT+QL+Text) compared to 8 arms that do not include Text (Control, BNI only, NRT only, QL only, BNI+NRT, BNI+QL, NRT+QL, BNI+NRT+QL); Test type: Superiority; p = 0.64, Regression, Logistic; adjusted for gender, age, race/ethnicity, baseline daily cigarette consumption; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.7 to 1.7]

ADVERSE EVENTS:
Time Frame: Each participant was monitored for adverse events for 3 months.
Arm/Group | NRT+QL+Text | BNI+QL+Text | BNI+NRT+QL+Text | NRT+QL | BNI+QL | NRT Only | BNI+Text | BNI+NRT+Text | NRT+Text | BNI+NRT | Control | BNI+NRT+QL | Text Only | QL+Text | BNI Only | QL Only
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 1/66 | 1/66 | 1/66
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/00/NCT02896400/Prot_SAP_000.pdf